CLINICAL TRIAL: NCT06978894
Title: Predicting Psychotic Relapse Using Speech-Based Early Detection
Acronym: MOTS+
Status: Recruiting | Type: Observational
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Lena Palaniyappan, Director, Centre of Excellence in Youth Mental Health, Douglas Mental Health University Institute
Other Study IDs: 2024-979
Record Dates: First submitted 2025-01-13; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-11

CONDITIONS: Psychosis
Keywords: psychosis; natural language processing; relapse; speech; relapse prediction
MeSH Terms: conditions — Psychotic Disorders; Recurrence; Speech

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Early Psychosis Patients: This study will participants recruited from three Early Psychosis Intervention (EPI) programs across Ontario and Quebec.
  This group will consist of approximately 250 patients experiencing or having experienced psychosis, enrolled in the EPI programs.

SUMMARY:
Psychotic disorders, including schizophrenia and affective psychosis, are severe mental health conditions marked by recurrent episodes that contribute to long-term disability. Relapses, characterized by the re-emergence of psychotic symptoms after remission, are a critical factor in the progression of these disorders, increasing risks such as suicide, cognitive impairment, and unemployment. This study aims to develop a novel, speech-based digital model to predict relapses in individuals with psychosis. Building on previous research into language abnormalities in schizophrenia, the study will employ a longitudinal design across Early Psychosis Intervention (EPI) clinics in Ontario and Quebec to advance relapse prediction

DETAILED DESCRIPTION:
OBJECTIVES: The primary goal of this study is to develop and validate a speech-based digital model to predict psychotic relapses in individuals with early psychosis. The study specifically aims to:

Test the hypothesis that within-subject changes in speech coherence, connectedness, and complexity, as measured by natural language processing (NLP) tools, will accurately identify imminent relapse, up to four weeks before clinical relapse in individuals receiving care in Early Psychosis Intervention (EPI) programs.

Investigate whether these speech-based relapse prediction models generalize across different languages (English and French) and are equally predictive in both males and females, addressing potential sociodemographic and linguistic influences on model performance.

Explore whether combining acoustic and prosodic features with core NLP-based speech measures improves the model's sensitivity and specificity for relapse prediction.

METHODS:

This study will employ a longitudinal, prospective design involving 250 first-episode psychosis (FEP) patients recruited from three Early Psychosis Intervention (EPI) clinics in Ontario and Quebec. The study aims to develop and evaluate a speech-based relapse prediction model, with a particular focus on generalizing results across different languages (English and French) and genders.

Participant Recruitment and Stratification:

Participants: A total of 250 FEP patients, including both English- and French-speaking individuals, will be enrolled to ensure linguistic diversity. The sample will be stratified by sex to evaluate model performance across genders.

Language groups: Approximately 60% of the participants will be English speakers and 40% French speakers, reflecting the population served by the EPI clinics.

Gender representation: The study aims to ensure that at least 40% of participants are female to assess gender-based differences in model prediction performance.

Baseline Assessments:

At baseline, participants will undergo a comprehensive in-person assessment to collect a detailed profile for each patient. This will include psychiatric symptomatology using the Positive and Negative Syndrome Scale (PANSS), Calgary Depression Scale and the Personal and Social Performance (PSP) scale, and cognitive functioning. Additionally, socioeconomic variables, historical and current medication usage, substance use (e.g., cannabis), and treatment adherence will also be recorded to provide a full clinical and treatment profile for each participant.

Speech Sampling and Data Collection:

Monthly Speech Samples: After the baseline assessment, participants will provide monthly speech samples over the course of 24 months. These speech samples will be collected using web-based prompts that include open-ended tasks, such as picture description or recall narratives, designed to elicit spontaneous speech.

Attrition and Speech Sample Estimates: Given an expected attrition rate of 35-50%, it is estimated that by the end of the study, 840-960 speech samples will be obtained from English-speaking participants and 660-870 speech samples from French-speaking participants.

Speech Analysis:

The collected speech samples will be analyzed using natural language processing (NLP) methods to extract key features associated with psychosis, including coherence (Measured by lexical predictability), Connectedness (Assessed using speech graph analysis) and Complexity (evaluated using the Analytic Thinking Index (ATI)). These NLP-derived speech metrics will be tracked over time to predict imminent psychotic relapses and compared across subgroups to assess the impact of language and gender on the predictive accuracy of the relapse model.

Data Analysis and Generalization:

The primary objective is to determine whether speech-based relapse prediction models generalize across different languages and genders. To achieve this, model performance will be evaluated across subgroups:

Linguistic subgroup analysis will compare the model's performance in English- and French-speaking participants.

Gender-based analysis will assess whether the predictive power of the speech-based model varies between male and female participants.

This analysis will ensure that the final model can be generalized across diverse populations and adapted for use in different clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age must be 16 years and older
* Diagnosis must meet DSM-5 criteria for psychotic disorders, including schizophrenia, schizoaffective disorder, or related conditions
* Fluency in English or French
* Must be currently receiving treatment through an EPI program

Exclusion Criteria:

* Severe comorbid speech or language disorders (e.g., aphasia)
* Primary diagnosis of non-psychotic disorders
* Inability to provide consent or complete assessments

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study population will consist of approximately 250 patients experiencing or having experienced psychosis, enrolled in the EPI programs.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Likelihood of relapse estimated using Speech-NLP Metrics | Monthly, up to 24 months
  This primary outcome will assess the ability of speech-based NLP metrics (coherence, connectedness, and complexity) to predict impending relapses in psychosis. Monthly speech samples will be analyzed to determine if changes in these metrics can distinguish timepoints preceding relapses from those not followed by relapse, with the aim of predicting relapses up to four weeks in advance. The likelihood of relapse is a numerical probabilistic estimate without any units. Outcome definition: Occurrence of relapse (i.e., psychiatric hospitalization, an increase in the level of psychiatric care, or substantial clinical deterioration >1wk that requires >25% increase in Defined Daily Dose equivalents of antipsychotics)
Generalization of Speech-Based Relapse Prediction Models Across Languages and Genders | Monthly, up to 24 months
  This outcome will assess whether the speech-based relapse prediction models are valid and perform equally well across different languages (English and French) and genders (male and female). The study will evaluate how sociodemographic factors such as language and sex impact the predictive accuracy of the models. NLP metrics (coherence, connectedness, complexity) will be correlated with clinical outcomes, and model performance will be compared across linguistic and gender subgroups to ensure generalizability.

SECONDARY OUTCOMES:
Likelihood of relapse estimated using multi-level speech features | Monthly, up to 24 months
  This exploratory outcome will assess the likelihood of relapse prediction by integrating acoustic features (e.g., speech rate, intonation), prosodic features (e.g., rhythm, pitch), and sentiment analysis into the primary measures (coherence, connectedness, complexity). Accuracy (the proportion of all relapse classifications that were correct, whether positive or negative) will be reported for the predictive models.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Robarts Research Institute, London, Ontario
  - Douglas Mental Health University Institute, Montreal, Quebec
  - Vitam, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
We propose to use a clinical linguistic archiving system called the TalkBank (https://www.talkbank.org/) for data sharing purposes. TalkBank registry/database is located at Carnegie Mellon University, Pittsburgh, Pennsylvania-USA. Several filters are used to de-identify the recorded speech data before storage in the databank. Firstly, the DISCOURSE protocol explicitly avoids using proper nouns and names/addresses. Second, the transcribed data is checked, and any proper names are replaced by common names (e.g., 'McGill' will be changed to 'University') or bleeped out (for audio data). If requested, we will play back the recorded responses to check if the participant is comfortable with the degree of anonymity. Identifying demographics will not be stored alongside the speech data to reduce triangulation. Finally, sharing is controlled by password protection, and a re-review is done to remove identifying information before sharing is initiated.
Supporting Information: Study Protocol
Time Frame: December 2028 for an unlimitied amount of time. There are no plans for data destruction of the study information stored (de-identified audio and transcriptions) within TalkBank.
Access Criteria: The anonymized speech data will be retained on an access-controlled secure database hosted by TalkBank.

REFERENCES:
- [Background] Zaher F, Diallo M, Achim AM, Joober R, Roy MA, Demers MF, Subramanian P, Lavigne KM, Lepage M, Gonzalez D, Zeljkovic I, Davis K, Mackinley M, Sabesan P, Lal S, Voppel A, Palaniyappan L. Speech markers to predict and prevent recurrent episodes of psychosis: A narrative overview and emerging opportunities. Schizophr Res. 2024 Apr;266:205-215. doi: 10.1016/j.schres.2024.02.036. Epub 2024 Feb 29. PMID 38428118